CLINICAL TRIAL: NCT00141908
Title: Prevention of Preterm Delivery in Twin Pregnancies by 17 Alpha-hydroxyprogesterone Caproate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Anwar Nassar, OB-GYN, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: OGY.AN.04
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Preterm Delivery
Keywords: Hydroxyprogesterone Caproate, twins, preterm delivery
MeSH Terms: conditions — Premature Birth | interventions — 17-alpha-Hydroxyprogesterone; 17 alpha-Hydroxyprogesterone Caproate; Castor Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo progesterone injection (Placebo Comparator): Placebo IM injections
  Interventions: Drug: Castor oil
- Progesterone injections (Active Comparator): 17-hydroxyprogesterone caproate weekly injections
  Interventions: Drug: 17-alpha Hydroxyprogesterone Caproate

INTERVENTIONS:
Drug: 17-alpha Hydroxyprogesterone Caproate — 250 mg IM weekly
  Other Names: Proluton depot
  Arms: Progesterone injections
Drug: Castor oil — weekly IM injections
  Arms: Placebo progesterone injection

SUMMARY:
Preterm birth remains a major cause of perinatal morbidity and mortality in developing as well as in developed countries. Despite major clinical research efforts aimed at reducing the incidence of preterm births in the United States, the preterm birth rate reached its highest level in 2 decades, 11.9% in 2001, which translates to a 27% rise since 1981. Much of this increase may be accounted for by the increase in multiple gestations brought about by assisted reproductive technology. Twin gestations accounting for 20% to 25% of all pregnancies conceived following such procedures. Twin gestations are at a particularly increased risk of preterm labor and they deliver at a mean gestational age of 37 weeks compared to 40 weeks for singleton pregnancies. In a study by our group, we estimated that about 54.5% of twin gestations would deliver prior to 37 completed weeks of gestation; i.e. preterm.

Evidence regarding efficacy of interventions designed to prevent preterm birth has been disappointing. Most well-designed clinical trials have failed to demonstrate any reduction in preterm births with such interventions as home uterine activity monitoring, reduced physical activity, administration of antibiotic or tocolytic therapy, and intensive and frequent antenatal follow ups. Recently, progesterone has shown some promise in the prevention of preterm birth among women with prior preterm births. Whether this intervention will prove effective in other populations, such as women with multiple gestations, remains to be seen.

The objective of our study is to compare the effectiveness of weekly intramuscular injections of 17-alpha Hydroxyprogesterone Caproate, a natural metabolite of progesterone, in preventing delivery at less than 37 weeks of gestation in a population of 290 patients with twin gestations between 16 and 36 weeks of gestation compared to a placebo. The data generated will be invaluable in managing this group of patients that is considered at a very high risk for preterm labor and delivery.

DETAILED DESCRIPTION:
Preterm birth remains the leading public health problem in obstetrics. A recent analysis of neonatal mortality (death at age < 28 days) in the United States between 1989 and 2001 revealed that preterm delivery (< 37 weeks) accounted for 70% of neonatal deaths.9 In addition to being at risk for neonatal death, preterm infants are at increased risk for long-term neurologic and developmental morbidity, with an estimated risk of significant handicaps in up to 15% of the survivors. These statistics have led many investigators to identify those women at greatest risk (e.g., those with prior preterm delivery, multiple gestations, maternal weight <50 kg, African-American race, bleeding, and concurrent sexually transmitted diseases). Despite identification of these risk factors, no reproducible and effective method of preventing preterm delivery has been demonstrated. On the contrary, preterm birth rates has risen 27% since 1981.1 A significant contributor to this tremendous rise is the increase in the rate of multiple gestations observed in over the past years. This is partly due to the advances in assisted reproductive technologies with twin gestations accounting for around a quarter of pregnancies conceived following these procedures.

One modality that showed promise for prevention of preterm labor in small trials was treatment with progestational agents. Two separate meta-analyses assessing the effects of progesterone on preterm labor arrived at contradictory conclusions. Goldstein found no evidence of effectiveness of progestational compounds in the prevention of preterm delivery. Daya, on the other hand, showed a beneficial effect. A third meta-analysis, restricted to trials of 17-alpha Hydroxyprogesterone Caproate showed, in composite, a significant reduction in the rate of preterm delivery. A recently reported trial comparing 17-alpha Hydroxyprogesterone Caproate therapy with placebo to prevent preterm birth in a select, high-risk group of women (documented history of a previous spontaneous preterm birth <37 weeks of gestation) was terminated prematurely when results showed a significant protection against recurrent preterm birth for women who received 17-alpha Hydroxyprogesterone Caproate. Other studies, using the same form of progesterone, did not demonstrate such a beneficial effect. A study in 1980 has failed to show any benefit of 17-alpha Hydroxyprogesterone Caproate in women with twin gestations. In that study, 77 women with twin gestations were treated during the last trimester with weekly injections of either 17-alpha Hydroxyprogesterone Caproate or a placebo. The study was limited by the small sample size. In addition, the progesterone therapy was started late in the third trimester of gestation which could partly explain the inability to detect a beneficial effect of progesterone in this group of patients using that particular regimen. Most reported trials on other progesterone compounds have failed to demonstrate a substantial effect in reducing the risk of preterm delivery. However, a recent small randomized placebo-controlled trial of supplemental vaginal progesterone in women at high risk for preterm birth revealed that the preterm birth rate at less than 34 weeks of gestation was significantly lower among women receiving progesterone than among those receiving placebo.8 The results of this study and that of the National Institute of Child Health and Human Development7 support the hypothesis that progesterone supplementation reduces preterm birth in a select very high-risk group of women. In fact, the American College of Obstetricians and Gynecologists Committee on Obstetric Practice believes that further studies are needed to evaluate the use of progesterone in patients with other high-risk obstetric factors, such as multiple gestations, short cervical length, or positive test results for cervicovaginal fetal fibronectin.

The mechanisms of action of 17-alpha Hydroxyprogesterone Caproate in prolonging gestation are not entirely known. They include relaxation of myometrial smooth muscle, blocking of the action of oxytocin, and inhibition of the formation of gap junctions. There is also evidence that local changes in the progesterone level or the ratio of progesterone to estrogen in the placenta, decidua, or fetal membranes may be important in the initiation of labor in humans. As for its safety profile, aside from local injection-site reactions like soreness, swelling, itching and bruising, 17-alpha Hydroxyprogesterone Caproate appears to be safe during pregnancy with absence of teratogenic effects. The safety of 17-alpha Hydroxyprogesterone Caproate administration in pregnancy is well documented by animal and clinical studies. Reviews of this topic by knowledgeable authors have uniformly concluded that no evidence exists that administration of 17-alpha Hydroxyprogesterone Caproate in pregnancy represents a significant risk to mother, fetus or newborn.

SPECIFIC AIM(S):

To test the effectiveness of weekly injections of 250 mg of 17-alpha Hydroxyprogesterone Caproate as compared with placebo in the prevention of preterm delivery in patients with twin gestations, when given from 16-20 weeks of gestation until 36 weeks.

We chose the 250 mg dose of 17-alpha Hydroxyprogesterone Caproate because this is the dose that was used in the studies that showed a beneficial effect of this medication in the prevention of preterm delivery.

The study hypothesis is that placebo is equivalent in its efficacy to 17-alpha Hydroxyprogesterone Caproate in preventing preterm delivery in twin pregnancies.

to participate in the trial.

Randomization procedure:

* We will stratify patients by reduced/non-reduced and IVF/ no-IVF. Patients will be then randomized to the different treatment groups using permuted block randomization.
* Randomization envelopes will be prepared by means of random number tables. Randomization will occur between 16 weeks and 20 weeks of gestation whereby the next numbered opaque envelope will be opened to assign each consenting patient to receive identically appearing active 17-alpha Hydroxyprogesterone Caproate (Proluton® Depot, Schering AG, Germany) or placebo (castor oil) injections prepared by our pharmacy.
* The women, their obstetricians, and research personnel will be blinded to the study medication allocation.
* A 2:1 ratio will be used for the assignment of women to 17-alpha Hydroxyprogesterone Caproate or placebo, because the patients assigned to placebo would be receiving painful injections on a weekly basis with no possibility of direct benefit.

Routine studies and procedures:

* An ultrasonographic examination, a routine procedure that is done on every pregnant patient, will be performed between 14 weeks and 20 weeks of gestation to confirm the gestational age and to identify any major fetal anomalies.
* Gestational age will be calculated based on the last menstrual period and/or first trimester ultrasonography for spontaneously conceived twins and the day of egg retrieval for twins conceived by assisted reproductive technology.

Interventions:

* After consenting, the patients will be offered to come for weekly injections of 17-alpha Hydroxyprogesterone Caproate (250 mg) or placebo given by a study nurse. If they cannot come for weekly injections, they will be handled the medications at the time of their follow up visits to their obstetricians to be given by a private nurse, whichever is more convenient for them. In order to avoid the burden on the clinic staff, it was decided to use the OPD premises from 11:30 a.m. to 1:30 p.m., a time where OPD sessions are over. Flow sheets to document the date of the injection will be available with the RA, obviating the need for pulling out patients charts. The financial compensation of the staff-nurse will comply with AUMBC rules and regulations.
* For those patients who elect to receive their injections at home, they will be called on the day of the injection to remind them of the injection to ensure that they are receiving the medication in due time.
* The patient will be categorized as non-compliant if there is ≥ 10 day-gap between any two injections.
* The injections will be continued until 36 weeks of gestation or delivery, whichever occurs first.
* In addition to the weekly visits for the study injections, the women will receive routine prenatal care with her obstetrician. Twin gestations at our department are usually asked to come for routine checkup visits every 3-4 weeks in the first and second trimester and every 2 weeks from 28 weeks to 36 weeks and weekly thereafter.
* The possible side effects of the medication, written in the consent form, will be explained to the patient by the research assistants.
* If a patient goes into preterm delivery, she will be managed by her obstetrician according to standard protocols that might necessitate admission and even tocolysis. In these cases, the injections will continue on a weekly basis till 36 weeks of gestation or delivery, whichever occurs first.

Statistical analysis Statistical analysis will be performed using the SPSS statistical package adjusting for the stratified design. The analyses will be done on the intent-to-treat basis. Categorical data like maternal characteristics and the rates of neonatal morbidity will be compared using Chi square when sample sizes support the approximation. Otherwise, categorical data will be analyzed with two-tailed Fisher exact test if the expected cell frequencies were small. Continuous variables will be compared by Student t test if assumptions of normality and homogeneity of variances appeared to be reasonable or the Wilcoxon rank-sum test. Unpaired variables and differences in distributions will be compared using the Mann-Whitney test. Neonatal outcomes will be analyzed on the assumption that if a neonatal outcome variable occurs in at least one of the fetuses, the pregnancy will be considered affected for that variable. A p-value <0.05 will be considered statistically significant.

A Logistic regression model will include all the confounding variables to for check their contribution to the primary outcome. The variables that we are going to control for include: need for tocolysis, BMI, smoking, assisted reproductive technology, prior preterm delivery, prior term delivery, spontaneous or reduced twins, etc ….

Prolongation of pregnancy will be assessed by life-table methods. The duration will be considered as the period between the time of randomization and the time a woman gives birth, is lost to follow-up, or reaches 40 weeks of gestation, whichever comes first.

CLINICAL RELEVANCE AND LIMITATIONS

* Managing preterm neonates is a major burden on the health system medically and financially. The results of this study will therefore have major implications if such treatment proves effective in reducing preterm delivery in twins.
* Limitations: Since the study is limited to twin gestations, the results cannot be generalized to singletons without risk factors for preterm labor or to higher order gestations.

ELIGIBILITY:
Inclusion Criteria:

* Viable twin pregnancy
* Current pregnancy between 16 weeks and 20 weeks of gestation

Exclusion Criteria:

* Known fetal anomaly in either twin
* Current or planned cervical cerclage
* Hypertension requiring medication
* Diabetes Mellitus
* Asthma
* History of deep vein thrombosis
* Preexisting cardiac or renal disease
* A seizure disorder
* Plans to deliver elsewhere
* Previous or existing liver tumors
* History of herpes gestationis of pregnancy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 290 (Estimated)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The frequency of delivery prior to completed 37 weeks of gestation (259 days). | one year

SECONDARY OUTCOMES:
Delivery before 35 weeks of gestation, Delivery before 32 weeks of gestation, Admission during current pregnancy for preterm labor, | 9 months
Need for tocolytic therapy in current pregnancy, Need for corticosteroids to enhance fetal lung maturity, Route of delivery, | 9 months
Obstetrical complications (antepartum and intrapartum) of pregnancy, Indicated preterm deliveries, Neonatal outcome variables ( Birth weight < 2500 grams, | 9 months
Birth weight < 1500 grams, Fetal death, antepartum or intrapartum, Neonatal intensive care unit admissions, Respiratory distress syndrome, | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Anwar H Nassar, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon